CLINICAL TRIAL: NCT01243307
Title: A Phase I, Single-centre, Multiple-dose, Placebo-controlled Crossover Study to Investigate the Pharmacodynamic Effects of CT327 (0.1% Topical Cream) on Intra-dermal Nerve Growth Factor (NGF) and Evoked Pain Responses, in Healthy Male Volunteers
Brief Title: A Study to Investigate the Pharmacodynamic Effects of CT327 on Intra-dermal Nerve Growth Factor (NGF) and Evoked Pain Responses, in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Creabilis SA (Industry)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Creabilis Therapeutics, Creabilis Therapeutics
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CT327-1002
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — pegcantratinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CT327 treatment period 1 (Experimental): Subjects in Group 1 will receive CT327 during treatment/testing period 1 and placebo during treatment/testing period 2
  Interventions: Drug: CT327 (or placebo) followed by placebo (or CT327)
- CT327 treatment period 2 (Experimental): Subjects in Group 2 will receive placebo during treatment/testing period 1 and CT327 during treatment/testing period 2
  Interventions: Drug: CT327 (or placebo) followed by placebo (or CT327)

INTERVENTIONS:
Drug: CT327 (or placebo) followed by placebo (or CT327) — During treatment/testing period 1, subjects will apply 0.25 g CT327 (or placebo) to 4 test fields of skin (2 on their arms and 2 on their legs) twice daily, 12 hours apart for a total of 7 applications.
  During treatment/testing period 2, subjects will apply 0.25 g placebo (or CT327) to 4 different test fields of skin (2 on their arms and 2 on their legs) twice daily, 12 hours apart for a total of 7 applications.

SUMMARY:
The primary objective of this study is to compare the effect of CT327 to placebo against experimental induced superficial, deep and hyperalgesic pain.

The secondary objectives are to elucidate the mechanisms of CT327 using experimental pain models.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to understand the contents of the study, comply with the study and willing to sign informed consent
* Subjects must be free from clinically significant illness or disease as determined by their medical history, physical examination, laboratory and other tests
* All male subjects must take adequate contraceptive precautions during the course of the study and for 30 days after their participation in the study has ended

Exclusion Criteria:

* Participation in other clinical studies within 3 months before screening
* Scheduled for surgery, medical treatment or any hospital admission that would fall within the study
* Use of strong painkillers
* Use of any analgesic within 24 hours before start of study
* Use of a regular course of prescribed medication and/or herbal medicine
* The presence of lesions, significant scars, cuts, wounds, dermal abnormalities, tattoos or naevi in the test areas
* A past history of contact dermatitis, psoriasis or keloid
* Any clinically significant ECG abnormality at screening
* A history of drug or other allergy that contraindicates his participation.
* Regular or average consumption of more than 21 units of alcohol per week (one unit of alcohol equals approximately 250 mL of beer, 125 mL of wine or 20 mL of spirits).
* Smokes more than five cigarettes (on average) per day, or had been a smoker of more than 5 cigarettes (on average) per day within the 3 months prior to screening.
* A known history of drug or alcohol abuse.
* As a result of the medical screening process, the PI or medical delegate considers the subject unfit for the study.
* Use of any prescription medication within 2 weeks or 5 half-lives (whichever is longer) of dosing.
* Use of non-prescription medication (e.g. aspirin, vitamins and herbal and dietary supplements) within 7 days prior to dosing, or 14 days if the medication contained grapefruit/ grapefruit juice or St John's Wort.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
An alteration in the peripheral sensitisation after treatment with CT327 | 2 treatment/testing periods each lasting 4 days and separated by at least 10 days

SECONDARY OUTCOMES:
The change in pain determined with the visual analogue scale (VAS) and the change in areas assessed with von Frey filaments and standardized brush. | 2 treatment/testing periods each lasting 4 days and separated by at least 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology Aalborg Hospital, Aalborg, Denmark